CLINICAL TRIAL: NCT00912106
Title: Boundary Lubrication of Synovial Fluid Molecules and Its Effect on the Surrounding Cells and Tissues
Brief Title: Analyzing Composition and Lubrication Properties of Synovial Fluid
Acronym: SFCL
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Science Concil (Unknown)
Responsible Party: Chih-Hung Chang, Division of Orthopedics, Far Eastern Memorial Hospital
Other Study IDs: 96024; NSC-96-
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Knee Osteoarthritis; HA Injection; One Injection Per Week for Five Week; Synovial Fluid Composition; Synovial Fluid Lubrication
Keywords: osteoarthritis; HA; synovial fluid; lubrication
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — synovial fluid from knee joint
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HA injection: Patients with osteoarthritis of knee. They are going to received HA injection 1 vial per week for 5 weeks.
  Interventions: Other: Synovial fluid composition and lubrication analysis

INTERVENTIONS:
Other: Synovial fluid composition and lubrication analysis — Before HA injection, synovial fluid must be drawn to increase treatment effectiveness. The drawn synovial fluid was then analyzed in the lab. There was no influence for patients enrolled because the drawn synovial fluid would usually be discarded.

SUMMARY:
To analyze the relationship between composition of synovial fluid and its lubrication properties

DETAILED DESCRIPTION:
Patients suffering from serious arthritis may receive the artificial joint replacement surgery. Comparing to the articulation of articular cartilage, the artificial joint undergo a boundary lubrication in which a thin layer of synovial fluid molecules is formed between the artificial joint materials. Therefore a larger wear rate is observed in the artificial joint system. Researchers have devoted themselves to modifying the artificial joint materials in order to reduce the wear phenomena. We first propose that modification the lubrication by adding effective lubricating molecules may help to reduce the wear of artificial joint. However, there still lacks fundamentally understanding of the artificial joint lubrication mechanism under synovial fluid. Hence, we plan to investigate the boundary lubrication mechanism of synovial molecules, such as albumin, globulin, hyaluronic acid, and lipid in the first year. We would like to obtain the adsorption behaviors of the single molecules as well as multiple molecules on the surfaces of artificial joint materials by experiments. Molecular dynamics simulation will also be performed to gain the knowledge of adsorption energy and possible conformation change of the molecules. In the second year, the tribological heat and mechanical effects on the synovial molecules will be studied. The analysis platform will be established to perform the composition and properties measurement of the synovial molecules. In the third year, we will further discuss the effect of the synovial molecules transformation on the surrounding cells and tissues. Their influences on the tribological and biochemical behaviors will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to receive HA injection of one or two knees

Exclusion Criteria:

* Patients whose quantity of synovial fluid is not enough to be drawn

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are going to receive HA injection of one or two knees
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Synovial fluid HA and albumin concentration; synovial fluid lubrication | 1 wk, 2 wk, 3 wk, 4 wk, 5 wk

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Chang, Ph. D, Study Director — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Pan-Ciao, Taipei, Taiwan